CLINICAL TRIAL: NCT00610818
Title: Effect of Palifermin Therapy on Benign and Malignant Skin Tumors in Patients Undergoing High-Dose Chemotherapy With Autologous Stem Cell Transplantation
Brief Title: Effect of Palifermin on Skin Tumors in Patients Undergoing Bone Marrow Transplantation
Acronym: Palifermin
Status: Terminated | Type: Observational
Why Stopped: We did not see any effect of Palifermin on benign or malignant tumor growth
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Dr. Beatrice Wang
Other Study IDs: BMB-6-24; BMB-06-24
Record Dates: First submitted 2008-01-28; First posted 2008-02-08 (Estimated); Last update posted 2008-02-08 (Estimated); Status verified 2008-01

CONDITIONS: Skin Rash
MeSH Terms: conditions — Exanthema | interventions — Fibroblast Growth Factor 7

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: Patients receiving palifermin to prevent mucositis from bone marrow transplant.
  Interventions: Other: Palifermin

INTERVENTIONS:
Other: Palifermin — day -14, -13, -12 before transplant and then day 0,1,2 after transplant
  Other Names: keratinocyte growth factor

SUMMARY:
We are approaching you to participate in this study because you are taking Palifermin and the purpose of this study is to describe the effect of Palifermin on skin growth found on the body. Palifermin is a new synthetic growth factor (encourages skin cells to grow) specifically designed to protect the areas of the body (mouth and upper digestive tract) that are damaged by chemotherapy. The cells in these areas are rapidly dividing cells and so are killed by chemotherapeutic drugs. Palifermin is a drug that stimulates new cells in these areas to grow and therefore protects patients from some serious side effects of chemotherapy. These include mucositis or inflammation of the lining of the mouth and other organs resulting in difficulty swallowing, speaking and extreme pain in the mouth and upper digestive tract.

Skin cells are also known to respond to these types of growth factors like Palifermin, but unfortunately no studies have been done that look specifically at the effect of this drug on pre-existing skin lesions or the development of new skin lesions. We will be asking you if you have noticed any change in moles or other skin lesions that you have, and if you have noticed any new lesions. We will also be doing a full physical examination of the skin at regular intervals during the study to document the appearance of any new lesions or change in pre-existing ones.

ELIGIBILITY:
Inclusion Criteria: receiving bone marrow transplant -

Exclusion Criteria: not receiving other growth factors

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients receiving palifermin for bone marrow transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2007-07; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: beatrice wang, MD, Principal Investigator — McGill University
Locations (1):
- McGill University, Montreal, Quebec, Canada